CLINICAL TRIAL: NCT03589066
Title: An Open-label, Randomized, Parallel-group Trial to Evaluate the Pharmacokinetics of Two Formulations of LY03003 After a Single Intramuscular Injection Administered to Patients With Parkinson's Disease
Brief Title: Pharmacokinetic Study of LY03003 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Luye Pharma Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY03003/CT-USA-104
Record Dates: First submitted 2018-06-08; First posted 2018-07-17 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Parkinson Disease
Keywords: rotigotine; parkinson; parkinsons; intramuscular injection; UPDRS
MeSH Terms: conditions — Parkinson Disease | interventions — rotigotine

STUDY DESIGN:
Intervention Model Description: Two different formulations of LY03003, i.e. Formulation A and Formulation B
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Formulation A (Experimental): LY03003 28 mg intramuscular suspension, single dose, 1 day duration
  Interventions: Drug: LY03003
- Formulation B (Experimental): LY03003 28 mg intramuscular suspension, single dose, 1 day duration
  Interventions: Drug: LY03003

INTERVENTIONS:
Drug: LY03003 — 28 mg intramuscular suspension
  Other Names: rotigotine

SUMMARY:
This is a Phase 1, open-label, parallel-group study to evaluate rotigotine pharmacokinetics, safety and tolerability following a single intramuscular dose of one of two different formulations of LY03003 in patients with Parkinson's disease.

DETAILED DESCRIPTION:
This study is designed to evaluate and compare the rotigotine pharmacokinetic profile of a single 28 mg intramuscular dose of LY03003 Formulation A and LY03003 Formulation B. The secondary objective of the trial is to evaluate the safety and tolerability of LY03003 Formulation A and LY03003 Formulation B following a single 28 mg IM dose administered to patients with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving informed consent and complying with trial procedures including the ability to stay at/return to the CRU for visits at the predetermined times on the prescribed schedule.
* Has idiopathic Parkinson's Disease (i.e., without any other known or suspected cause of Parkinsonism) defined by the cardinal signs, bradykinesia, plus the presence of ≥1 of the following: resting tremor, rigidity, or impairment of postural reflexes.
* Male or female patient ≥18 years old with BMI of 18.5 to 32 kg/m2, inclusive, and body weight ≥50 kg at Screening.
* MMSE score ≥25 at Screening.
* UPDRS motor (Part III) score ≥ 10 but ≤ 42 at Screening.
* All female patients (childbearing potential and non-childbearing potential) must have a negative serum pregnancy test result at Screening. In addition, female patients must meet 1 of the following 3 conditions: (i) postmenopausal for at least 12 months without an alternative medical cause, (ii) surgically sterile (hysterectomy, bilateral oophorectomy, bilateral salpingectomy, or bilateral tubal occlusion) based on patient report, or (iii) if of childbearing potential, practicing or agree to practice a highly effective method of contraception.

Exclusion Criteria:

* Atypical Parkinson's syndrome(s) due to drugs (e.g., metoclopramide, flunarizine), metabolic neurogenetic disorders (e.g., Wilson's Disease), encephalitis, cerebrovascular disease, or degenerative disease (e.g., progressive Supranuclear Palsy).
* History of pallidotomy, thalamotomy, deep brain stimulation, or fetal tissue transplant.
* Dementia, active psychosis or hallucinations, or clinically significant major depression requiring psychiatric interventions.
* Lifetime history of suicide attempt (including an active attempt, interrupted attempt, or aborted attempt) or suicidal ideation in the past 6 months as indicated by a positive response ("Yes") to either Question 4 or Question 5 of the C-SSRS.
* History of symptomatic orthostatic hypotension with a decrease of ≥20 mmHg in SBP or decrease of ≥10 mmHg in DBP when changing from supine to standing position after having been in the supine position for at least 5 minutes or SBP less than 105 mmHg in a supine position at the Screening Visit.
* Therapy with a dopamine (DA) agonist either concurrently or within 21 days prior to study drug dosing.
* Therapy with 1 or more of the following drugs either concurrently or within 21 days prior to study drug dosing: monoamine oxidase inhibitors, DA releasing agents, DA modulating agents, DA antagonists, DA depleting antihypertensives, tricyclic antidepressants, neuroleptics, or other medications that may interact with DA function.
* Current diagnosis of epilepsy, history of seizures as an adult, lifetime history of stroke, or transient ischemic attack (TIA) within 1 year prior to the Screening Visit.
* Female patient who is pregnant or breastfeeding or of childbearing potential without adequate contraception
* History of prescription drug abuse or illicit drug use, alcohol abuse, or tobacco use within 6 months prior to the Screening Visit or positive finding in drugs of abuse test, nicotine test, or alcohol test.
* Any other clinically relevant hepatic, renal, hematologic, and/or cardiac dysfunction, or other medical condition, or clinically significant laboratory abnormality that would interfere with the patient's safety or trial outcome in the judgment of the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Cmax | 22 days
  Maximum plasma concentration
AUClast | 22 days
  Area under the concentration-time curve up to the time of the last measurable concentration
AUCinf | 22 days
  Area under the concentration-time curve from time zero extrapolated to infinity

SECONDARY OUTCOMES:
Frequency of adverse events | screening, baseline and days 1, 2, 3, 5, 7, 9, 12, 15, 18 and Day 22
  Adverse events
Frequency of serious adverse events | screening, baseline and days 1, 2, 3, 5, 7, 9, 12, 15, 18 and Day 22
  Serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Booth, MD, DVM, Study Director — Luye Pharma Group Ltd.
Locations (2):
- United States (2):
  - MD Clinical, Hallandale, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No